CLINICAL TRIAL: NCT00982137
Title: Randomised, Double-blind, Phase II Evaluation of the Safety and Immunogenicity Following Administration of Live Attenuated JE Vaccine (ChimeriVax™-JE) and Yellow Fever Vaccine (STAMARIL®)
Brief Title: Study of Live Attenuated Japanese Encephalitis Vaccine (ChimeriVax™-JE) and Yellow Fever Vaccine (STAMARIL®)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-006
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Japanese Encephalitis; Yellow Fever
Keywords: Japanese Encephalitis; Yellow Fever; ChimeriVax™-JE; STAMARIL®; Adult
MeSH Terms: conditions — Encephalitis, Japanese; Yellow Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ChimeriVax™-JE then STAMARIL® (Experimental): Participants will receive ChimeriVax™-JE on Day 0 and STAMARIL® on Day 30
  Interventions: Biological: Live attenuated Japanese encephalitis virus; Yellow fever virus
- STAMARIL® then ChimeriVax™-JE (Experimental): Participants will receive STAMARIL® on Day 0 and ChimeriVax™-JE on Day 30
  Interventions: Biological: Yellow fever virus; Live attenuated Japanese encephalitis virus
- ChimeriVax™-JE and STAMARIL®, then Diluent (Experimental): Participants will receive ChimeriVax™-JE and STAMARIL® on Day 0 and diluent on Day 30.
  Interventions: Biological: Live attenuated Japanese encephalitis virus; Yellow fever virus
- Diluent then ChimeriVax™-JE and STAMARIL® (Experimental): Participants will receive Diluent on Day 0 and ChimeriVax™-JE and STAMARIL® on Day 30.
  Interventions: Biological: Live attenuated Japanese encephalitis virus; Yellow fever virus

INTERVENTIONS:
Biological: Live attenuated Japanese encephalitis virus; Yellow fever virus — ChimeriVax™-JE, 0.5 mL, Subcutaneous on Day 0; STAMARIL®, 0.5 mL, Subcutaneous on Day 30.
  Other Names: ChimeriVax-JE; STAMARIL®
  Arms: ChimeriVax™-JE then STAMARIL®
Biological: Yellow fever virus; Live attenuated Japanese encephalitis virus — STAMARIL®, 0.5 mL Subcutaneous on Day 0; ChimeriVax™-JE, 0.5 mL Subcutaneous on Day 30.
  Other Names: STAMARIL®; ChimeriVax™-JE
  Arms: STAMARIL® then ChimeriVax™-JE
Biological: Live attenuated Japanese encephalitis virus; Yellow fever virus — ChimeriVax™-JE, 0.5 mL Subcutaneous and STAMARIL®, 0.5 mL, Subcutaneous on Day 0; Diluent 0.5 mL, Subcutaneous on Day 30.
  Other Names: ChimeriVax™-JE; STAMARIL®
  Arms: ChimeriVax™-JE and STAMARIL®, then Diluent
Biological: Live attenuated Japanese encephalitis virus; Yellow fever virus — Diluent, 0.5 mL Subcutaneous on Day 0; ChimeriVax™-JE, 0.5 mL Subcutaneous and STAMARIL®, 0.5 mL Subcutaneous on Day 30.
  Other Names: ChimeriVax™-JE; STAMARIL®
  Arms: Diluent then ChimeriVax™-JE and STAMARIL®

SUMMARY:
The purpose of this study is to obtain safety, tolerability, and immunogenicity data on the co-administration or sequential administration of Chimeravax™-JE vaccine and STAMARIL®.

Objectives:

Safety:

* Obtain safety and tolerability data of a single, fixed dose of ChimeriVax™-JE administered concurrently, one month before or one month after STAMARIL® to adult volunteers (≥ 18 to ≤ 55 years) without prior Japanese encephalitis (JE) or yellow fever (YF) vaccination.

Immunogenicity:

* Obtain data on the antibody response to a single, fixed dose of ChimeriVax™-JE administered concurrently, one month before or one month after STAMARIL® to adult volunteers without prior JE (or YF) vaccination.
* Assess the durability of the immune response in adult volunteers 6 months after administration of ChimeriVax™-JE and STAMARIL®.

DETAILED DESCRIPTION:
All participants will receive two injections, one to each arm on Days 0 and 30, respectively. Immunogenicity will be tested on Days 0, 15, 30, 45, and 60, and at Month 6.

ELIGIBILITY:
Inclusion Criteria :

* All aspects of the protocol explained and written informed consent obtained from the participant.
* Aged ≥ 18 to ≤ 55 years at Day 0.
* In good general health, without significant medical history, physical examination findings, or clinically significant abnormal laboratory results.
* Participant must be available for the study duration, including all planned follow-up visits.
* The participant must agree to take the following precautions to avoid insect bites for 7 days following vaccination: (a) wear long-sleeved shirts and trousers; (b) apply N,N-Diethyl-meta-toluamide (DEET)-containing insect repellents; (c) sleep in screened enclosures.
* Female participants of childbearing potential must have a negative serum pregnancy test. An efficacious hormonal method (i.e., oral, implantable or injectable) of contraception or an intrauterine contraceptive device (IUCD) must be used at least 1 month before Screening and at least 1 month after Day 60. These participants will sign an agreement that contraception will be practised during the specified periods and will specify the method used. Female participants unable to become pregnant must have this documented (e.g., tubal ligation or hysterectomy).

Exclusion Criteria :

* A history of flavivirus infection or vaccination to Japanese encephalitis (JE) or yellow fever (YF). Previous vaccination will be determined by history (interview of subject) and/or by reviewing the participant's vaccination card or other official documentation (either a history of or documentation of vaccination fulfils the criterion for exclusion).
* Impaired immunity, including known or suspected immunodeficiency (e.g., human immunodeficiency virus [HIV] infection, primary immunodeficiency disorder, leukemia, lymphoma), use of immunosuppressive or antineoplastic drugs (including corticosteroids > 10 mg prednisone, or equivalent, for more than 14 days in the last three months).
* Clinically significant abnormal laboratory assessment results.
* Serious adverse reactions characterised by urticaria or angioedema to a prior vaccine, chicken or eggs or egg protein.
* Transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin, within six months of the Screening Visit or up to Day 60.
* Administration of another vaccine within 28 days of receiving study vaccination.
* Physical examination indicating any clinically significant medical condition including any short-lived or long-standing illness which has become more severe.
* Body temperature >38.1°C (100.6°F) or acute illness within 3 days prior to inoculation (participant may be rescheduled).
* Intention to travel out of the area prior to the study visit on Day 60.
* Seropositive to hepatitis C virus (HCV) or HIV or positive for hepatitis B virus (HBV) (antigen).
* Lactation or intended pregnancy in female participants.
* Excessive alcohol consumption, drug abuse, significant psychiatric illness.
* A known or suspected physiological or structural condition that compromises the integrity of the blood-brain barrier (e.g., significant hypertensive cerebrovascular disease, trauma, ischaemia, infection, inflammation of the brain).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2004-07; Primary Completion 2005-04 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Herston, Queensland, Australia

REFERENCES:
- [Result] Nasveld PE, Marjason J, Bennett S, Aaskov J, Elliott S, McCarthy K, Kanesa-Thasan N, Feroldi E, Reid M. Concomitant or sequential administration of live attenuated Japanese encephalitis chimeric virus vaccine and yellow fever 17D vaccine: randomized double-blind phase II evaluation of safety and immunogenicity. Hum Vaccin. 2010 Nov;6(11):906-14. doi: 10.4161/hv.6.11.12854. Epub 2010 Nov 1. PMID 20864814
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled from 27 July 2004 to 27 September 2004 at 1 clinical center in Australia.
Pre-assignment Details: A total of 108 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- ChimeriVax™-JE Then STAMARIL®: All participants received a single ChimeriVax™-JE vaccine on Day 0 and a single dose of STAMARIL® vaccine on Day 30.
- STAMARIL® Then ChimeriVax™-JE: All participants received a single dose of STAMARIL® vaccine on Day 0 and a single dose of ChimeriVax™-JE vaccine on Day 30.
- Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent: All participants received 1 dose each of ChimeriVax™-JE (left arm) and STAMARIL® (right arm) on Day 0 and diluent in the left and right arms on Day 30.
- Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®: All participants received diluent vaccination (left and right arms)on Day 0, followed with STAMARIL® (left arm) and ChimeriVax™-JE (right arm) on Day 30.
Period: Overall Study
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Started | 36 | 36 | 18 | 18
Completed | 36 | 35 | 18 | 17
Not Completed | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL® | Total
Number analyzed (Participants) | 36 | 36 | 18 | 18 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 18 | 18 | 108
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 27.2 (9.71) | 23.4 (6.95) | 27.5 (10.19) | 25.8 (8.26) | 25.8 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 10 | 7 | 46
  Male | 20 | 23 | 8 | 11 | 62
Region of Enrollment [Number; unit: Participants]
  Australia | 36 | 36 | 18 | 18 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Japanese Encephalitis Seroconversion Following ChimeriVax™-JE or STAMARIL® Alone or the Co-administration of ChimeriVax™-JE and STAMARIL®, or Placebo Vaccination.
Description: Neutralising antibody titer against homologous Japanese encephalitis (JE), yellow fever (YF), and other relevant wild type JE strains were determined using a 50% serum dilution plaque reduction neutralisation test. Seroconversion post-vaccination was defined as the appearance of neutralising antibody titer when not present at Day 0, or at least a four-fold rise in neutralising antibody titer between the pre-vaccination (Day 0) and the post-vaccination samples.
  The 30 Days post-JE seroconversion is: Day 30 for Group 1 (ChimeriVax™-JE then STAMARIL®) and Group 3 (Co-administration of ChimeriVax™-JE and STAMARIL, then Diluent); Day 60 for Group 2 (STAMARIL® then ChimeriVax™-JE) and Group 4 (Diluent then Co-administration of ChimeriVax™-JE and STAMARIL).
Time Frame: Pre-vaccination (Day 0 or 30) and post-vaccination (Day 30 or 60)
Population: Japanese encephalitis seroconversion was assessed in all participants who were flavivirus naive at Day 0 and who had no protocol violations that might have interfered with analysis of primary endpoints (Per-Protocol Population).
Measure: Number; unit: Participants
Groups:
- ChimeriVax™-JE Then STAMARIL®: Participants received a single ChimeriVax™-JE on Day 0 and a single dose of STAMARIL® on Day 30.
- STAMARIL® Then ChimeriVax™-JE: Participants received a single dose of STAMARIL® on Day 0 and a single dose of ChimeriVax™-J on Day 30.
- Co-administration of ChimeriVax™-JE and STAMARIL, Then Diluent: Participants received 1 dose each of ChimeriVax™-JE (left arm) and STAMARIL® (right arm) on Day 0 and diluent in both left and right arms on Day 30.
- Diluent Then Coadministration With ChimeriVax™-JE and STAMARIL: Subjects received sc vaccination with diluent (both left and right arms) on Day 0, then sc vaccination with ChimeriVax™-JE (right arm) and STAMARIL® (left arm) on Day 30.
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL, Then Diluent | Diluent Then Coadministration With ChimeriVax™-JE and STAMARIL
Number analyzed (Participants) | 17 | 23 | 13 | 10
Participants
  Day 30 (N = 17, 23, 13, 10) | 17 | 2 [0 to 0] | 12 | 0
  Day 60 (N = 17, 23, 13, 10) | 17 | 21 | 12 | 10
  30 Days Post-JE Seroconversion (N = 17, 23, 23, 0) | 17 | 21 | 22 | NA — Data for the participants in Group 3 (Co-administration of ChimeriVax™-JE and STAMARIL®, then Diluent) and Group 4, (Diluent then co-administration with ChimeriVax™-JE and STAMARIL) were pooled and presented in Group 3 column.

2. Primary Outcome: Number of Participants With Yellow Fever Seroconversion Following ChimeriVax™-JE or STAMARIL® Alone or the Co-administration of ChimeriVax™-JE and STAMARIL® or Placebo Vaccination.
Description: Neutralising antibody titer against yellow fever strains was determined using a 50% serum dilution plaque reduction neutralisation test. Seroconversion at a later post vaccination timepoint ws defined as the appearance of neutralising antibody titer when not present at Day 0, or at least a four-fold rise in neutralising antibody titre between the pre-injection Day 0 and later post vaccination samples.
  The Day 30 post-JE seroconversion is: Day 30 for Group 1 (ChimeriVax™-JE then STAMARIL®) and Group 3 (Co-administration of ChimeriVax™-JE and STAMARIL, then Diluent); Day 60 for Group 2 (STAMARIL® then ChimeriVax™-JE) and Group 4 (Diluent then Co-administration of ChimeriVax™-JE and STAMARIL).
Time Frame: Pre-vaccination (Day 0 or 30) and post-vaccination (Day 30 or 60)
Population: Yellow fever seroconversion was assessed in all participants who were flavivirus naive at Day 0 and who had no protocol violations that might have interfered with analysis of primary endpoints (Per Protocol Population).
Measure: Number; unit: Participants
Groups:
- Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent: Participants received 1 dose each of ChimeriVax™-JE (left arm) and STAMARIL® (right arm) on Day 0 and diluent in both left and right arms on Day 30.
- Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®: Subjects received STAMARIL® then ChimeriVaxTM-JE vaccination with diluent (both left and right arms) on Day 0, then STAMARIL® then ChimeriVaxTM-JE vaccination with ChimeriVax™-JE (right arm) and STAMARIL® (left arm) on Day 30.
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Number analyzed (Participants) | 17 | 23 | 13 | 10
Participants
  Day 30 (N = 17, 23, 13, 10) | 0 | 23 | 13 | 1
  Day 60 (N = 17, 23, 13, 10) | 17 | 23 | 13 | 10
  Day 30 Post-JE Seroconversion (N = 17, 23, 23, 0) | 17 | 23 | 23 | NA — Data for the participants in Group 3 (Co-administration of ChimeriVax™-JE and STAMARIL, then Diluent) and Group 4, (Diluent then co-administration with ChimeriVax™-JE and STAMARIL) were pooled and presented in Group 3 column.

3. Secondary Outcome: Geometric Mean Titers (GMTs) to Japanese Encephalitis (Homologous Virus) Following ChimeriVax™-JE or STAMARIL® Alone or the Co-administration of ChimeriVax™-JE and STAMARIL®, or Placebo Vaccination.
Description: Neutralising antibody titer against homologous Japanese encephalitis (JE) and other relevant wild type JE strains was determined using a 50% serum dilution plaque reduction neutralisation test.
  Post-vaccination 15 (30) Days JE seroconversion is: Day 15 (30) for Group 1 (ChimeriVax™-JE then STAMARIL®) and Group 3 (Co-administration of ChimeriVax™-JE and STAMARIL, then Diluent); Day 45 (60) for Group 2 (STAMARIL® then ChimeriVax™-JE) and Group 4 (Diluent then Co-administration of ChimeriVax™-JE and STAMARIL)
Time Frame: Day 0 through 6 months post-vaccination
Population: GMTs were assessed in all participants who were flavivirus naive at Day 0 and who had no protocol violations that might have interfered with analysis of primary endpoints (Per-protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Number analyzed (Participants) | 17 | 23 | 13 | 10
Titers
  15 Days Post-vaccination (N = 17, 23, 13, 10) | 282.1 [130.8 to 608.3] | 140.2 [50.9 to 386.3] | 119.9 [53.6 to 267.9] | 386.5 [135.1 to 1106.4]
  30 Days Post-vaccination (N = 17, 23, 13, 10) | 1461.6 [632.8 to 3375.8] | 426.4 [172.3 to 1055.1] | 221.2 [94.9 to 515.3] | 611.6 [188.4 to 1986.0]
  45 Days Post-vaccination (N = 17, 0, 13, 0) | 1099.3 [465.9 to 2593.6] | NA [NA to NA] — Data were not assessed at this time point for this group. | 146.3 [58.3 to 367.2] | NA [NA to NA] — Data were not assessed at this time point for this group.
  60 Days Post-vaccination (N = 17, 0, 13, 0) | 687.8 [315.4 to 1499.8] | NA [NA to NA] — Data were not assessed at this time point for this group. | 103.1 [43.9 to 242.1] | NA [NA to NA] — Data were not assessed at this time point for this group.
  6 Months Post-vaccination (N = 16, 22, 13, 10) | 267.5 [122.4 to 584.4] | 134.0 [59.2 to 303.4] | 94.6 [37.8 to 236.9] | 99.9 [56.8 to 175.7]

4. Secondary Outcome: Geometric Mean Titers to Yellow Fever (Homologous Virus) Following ChimeriVax™-JE or STAMARIL® Alone or the Co-administration of ChimeriVax™-JE and STAMARIL®, or Placebo
Description: Neutralising antibody titer against homologous yellow fever was determined using a 50% serum dilution plaque reduction neutralisation test.
  Post vaccination 15 (30) Days Yellow Fever seroconversion is: Day 15 (30) for Group 1 (ChimeriVax™-JE then STAMARIL®) and Group 3 (Co-administration of ChimeriVax™-JE and STAMARIL, then Diluent); Day 45 (60) for Group 2 (STAMARIL® then ChimeriVax™-JE) and Group 4 (Diluent then Co-administration of ChimeriVax™-JE and STAMARIL).
Time Frame: Day 0 through 6 months post-vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Number analyzed (Participants) | 17 | 23 | 13 | 10
Titers
  Day 15 Post-vaccination (N = 17, 23, 13, 10) | 463.1 [156.2 to 1372.8] | 1080.7 [606.3 to 1926.2] | 1150.0 [527.3 to 2507.8] | 2044.1 [768.7 to 5435.2]
  Day 30 Post-vaccination (N = 17, 23, 13, 10) | 3288.5 [1415.4 to 7640.4] | 3704.6 [2271.4 to 6042.0] | 1565.6 [897.9 to 2729.9] | 3054.9 [1230.2 to 7586.3]
  Day 45 Post-vaccination (N = 0, 23, 13, 0) | NA [NA to NA] — Data were not assessed at this time point for this group. | 2442.5 [1450.5 to 4112.8] | 974.6 [572.3 to 1659.8] | NA [NA to NA] — Data were not assessed at this time point for this group.
  Day 60 Post-vaccination (N = 0, 23, 13, 0) | NA [NA to NA] — Data were not assessed at this time point for this group. | 2175.1 [1223.9 to 3865.4] | 653.1 [277.2 to 1539.0] | NA [NA to NA] — Data were not assessed at this time point for this group.
  6 Months Post-vaccination (N = 16, 22, 13, 10) | 2017.5 [842.0 to 4834.3] | 2058.7 [1302.5 to 3253.8] | 947.4 [431.3 to 2081.3] | 1351.8 [534.9 to 3416.4]

5. Primary Outcome: Number of Participants Who Seroconverted to Japanese Encephalitis 30 Days Post ChimeriVax™-JE Vaccination
Description: Neutralising antibody titer against homologous JE, YF, and other relevant wild type JE strains was determined using a 50% serum dilution plaque reduction neutralisation test. Seroconversion at a later post vaccination timepoint was defined as the appearance of neutralising antibody titer when not present at Day 0, or at least a four-fold rise in neutralising antibody titer between the pre-injection Day 0 and post-vaccination samples.
Time Frame: Day 0 (Pre-vaccination) through Day 30 post-vaccination
Population: Japanese encephalitis seroconversion was assessed in all participants who were flavivirus naive at Day 0 and who had no protocol violations that might have interfered with analysis of primary endpoints (Per Protocol Population).
Measure: Number; unit: Participants
Groups:
- STAMARIL® Then ChimeriVax™-JE: Participants received a single dose of STAMARIL® on Day 0 and a single dose of ChimeriVax™-JE on Day 30.
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Number analyzed (Participants) | 17 | 23 | 13 | 10
Participants
  JE Homologous Virus | 17 | 21 | 12 | 10
  Genotype I | 17 | 21 | 13 | 10
  Genotype II | 15 | 16 | 9 | 9
  Genotype III | 16 | 20 | 9 | 10
  Genotype IV | 15 | 15 | 5 | 9

6. Primary Outcome: Number of Participants Reporting Solicited Local and Systemic Adverse Events Post Vaccination With ChimeriVax™-JE or STAMARIL® Alone or the Co-Administration of ChimeriVax™-JE and STAMARIL®, or Placebo
Description: Solicited Local Adverse Events: Injection Site Pain, Erythema, Swelling, Hemorrhage, Venipuncture site Hemorrhage. Solicited Systemic Adverse Events: Fatigue, Malaise, Pyrexia, Chills, Headache, Dizziness, Myalgia, Abdominal Pain, Diarrhea, Nausea, Pharyngolaryngeal Pain.
  All solicited local reactions associated with ChimeriVax™-JE are presented in Group 1, those associated with STAMARIL® in Group 2, those associated with co-administered vaccines in Group 3, and those associated with diluent in Group 4. The solicited systemic adverse events are reported according to the participants' randomized study groups.
Time Frame: Day 0 up to Day 60 post-vaccination
Population: Safety analyses were performed on data from all randomized subjects who received at least one dose of study medication: ChimeriVax JE, STAMARIL, or Diluent (Safety Population).
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Number analyzed (Participants) | 71 | 72 | 36 | 36
Participants
  Injection Site Pain (N = 71, 72, 36, 36) | 13 | 13 | 6 | 4
  Injection Site Erythema (N = 71, 72, 36, 36) | 6 | 9 | 3 | 1
  Injection Site Swelling (N = 71, 72, 36, 36) | 4 | 0 | 3 | 1
  Injection Site Hemorrhage (N = 71, 72, 36, 36) | 1 | 2 | 1 | 0
  Venipuncture Site Hemorrhage (N = 71, 72, 36, 36) | 0 | 2 | 0 | 0
  Fatigue (N = 36, 36, 18, 18) | 16 | 15 | 3 | 10
  Malaise (N = 36, 36, 18, 18) | 10 | 12 | 2 | 6
  Pyrexia (N = 36, 36, 18, 18) | 3 | 4 | 0 | 3
  Chills (N = 36, 36, 18, 18) | 1 | 4 | 1 | 2
  Headache (N = 36, 36, 18, 18) | 18 | 20 | 6 | 8
  Dizziness (N = 36, 36, 18, 18) | 0 | 2 | 0 | 0
  Myalgia (N = 36, 36, 18, 18) | 7 | 12 | 3 | 4
  Abdominal Pain (N = 36, 36, 18, 18) | 5 | 4 | 2 | 3
  Diarrhea (N = 36, 36, 18, 18) | 7 | 2 | 2 | 3
  Nausea (N = 36, 36, 18, 18) | 3 | 1 | 1 | 2
  Pharyngolaryngeal Pain (N = 36, 36, 18, 18) | 0 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0, after vaccination up to Month 6 post-vaccination.
Description: Solicited local reactions associated with ChimeriVax™-JE are presented in Group 1; associated with STAMARIL® in Group 2; associated co-administered vaccines in Group 3, and associated with diluents in Group 4. Solicited systemic reactions and unsolicited adverse events are reported according to the participants' randomized study groups.
Arm/Group | ChimeriVax™-JE Then STAMARIL® | STAMARIL® Then ChimeriVax™-JE | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL®
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 18/71 | 20/72 | 6/36 | 10/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ChimeriVax™-JE Then STAMARIL® (N=71) | STAMARIL® Then ChimeriVax™-JE (N=72) | Co-administration of ChimeriVax™-JE and STAMARIL® Then Diluent (N=36) | Diluent Then Coadministration With ChimeriVax-JE and STAMARIL® (N=36)
Fatigue (General disorders) | 16/36 | 15/36 | 3/18 | 10/18
Injection Site Pain (General disorders) | 13 | 13 | 6 | 4
Injection Site Erythema (General disorders) | 6 | 9 | 3 | 1
Injection Site Swelling (General disorders) | 4 | 0 | 3 | 1
Malaise (General disorders) | 10/36 | 12/36 | 2/18 | 6/18
Pyrexia (General disorders) | 3/36 | 4/36 | 0/18 | 3/18
Chills (General disorders) | 1/36 | 4/36 | 1/18 | 2/18
Headache (Nervous system disorders) | 18/36 | 20/36 | 6/18 | 8/18
Dizziness (Nervous system disorders) | 0/36 | 2/36 | 0/18 | 0/18
Myalgia (Musculoskeletal and connective tissue disorders) | 7/36 | 12/36 | 3/18 | 4/18
Abdominal Pain (Gastrointestinal disorders) | 5/36 | 4/36 | 2/18 | 3/18
Diarrhea (Gastrointestinal disorders) | 7/36 | 2/36 | 2/18 | 3/18
Nausea (Gastrointestinal disorders) | 3/36 | 1/36 | 1/18 | 2/18
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0/36 | 2/36 | 0/18 | 1/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.